CLINICAL TRIAL: NCT02156479
Title: Clinical Validation of an Improved T-Track® CMV Assay to Assess the Functionality of CMV Protein-reactive Cell-mediated Immunity (CMI) and Its Suitability to Determine a Protective Cut-off Value for Recurrent CMV Reactivations in Allo-HSCT Recipients
Brief Title: Clinical Validation of Lophius Biosciences Kit T-Track® CMV in Allo-HSCT Recipients
Acronym: AlloProtectCMV
Status: Completed | Type: Observational
Sponsor: Lophius Biosciences GmbH (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: LB-B1
Record Dates: First submitted 2014-05-27; First posted 2014-06-05 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Cytomegalovirus Infection; GVHD
Keywords: CMV; T-Track CMV; allo-HSCT; CMI
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Allo-HSCT recipients: Patients receiving an allogeneic hematopoietic stem cell transplantation for the first time, being either CMV seropositive or receiving a graft from a CMV seropositive donor or both, donor and recipient are CMV seropositive

SUMMARY:
This study in a cohort of allo-HSCT recipients aims to validate the suitability of an improved T-Track® CMV assay to assess the functionality of CMV protein-reactive effector cells and its suitability to determine cut-off values mediating protection from recurrent CMV reactivations in allo-HSCT recipients.

Lophius T-Track® CMV represents a highly standardized and sensitive diagnostic tool to assess the functionality of a network of clinically relevant CMV-reactive effector cells. It is based on the stimulation of peripheral blood mononuclear cells (PBMC) with activated immunodominant CMV proteins, pp65 and IE-1, and the subsequent quantification of CMV-specific CMI (spot forming colonies) using a highly sensitive IFN-γ ELISpot.

DETAILED DESCRIPTION:
CMV reactivation after allogeneic hematopoietic stem cell transplantation (allo-HSCT) is associated with significant morbidity and increased overall mortality. Patients are generally pre-emptively treated with antiviral medication after elevated levels of CMV copies in peripheral blood or plasma have been detected by quantitative PCR. However, these CMV reactivations are often subclinical and do not lead to complications or CMV disease. In these cases functional CMV- specific effector cells have been shown to mediate protection from clinical symptoms. Monitoring of CMV- specific effector cells after allo-HSCT could help to prevent severe side effects due to unnecessary antiviral treatment.

Since the majority of patients develops more than one episode of CMV reactivation, determination of functional CMV-reactive effector cells of cell mediated immunity (CMI) could also help to predict the likelihood of relapsing CMV reactivations and thereby adjust the need for and duration of secondary prophylaxis.

Currently available techniques to measure CMV-specific effector cells lack either a functional read out (multimer stain) or are time consuming and difficult to standardize (detection of intracellular interferon gamma (IFN-ᵞ) after in vitro stimulation using flow cytometry). The improved T-Track® CMV assay has the advantage of combining a standardized and highly sensitive test system with a functional read out (IFN-ᵞ production) considering the function of antigen presenting cells (APC) and different populations of clinically relevant effector cells (CTL, T helper-, NK-, NKT cells). Based on experiences of the performance of this assay system in healthy individuals and hemodialysis patients (the latter as part of a performance evaluation - EUDAMED number 00015561) the presented trial aims to validate an improved variant of this test (including optimized, LPS-depleted IE-1 protein) with regard to its suitability to predict freedom from relapse of CMV-reactivation following treatment of CMV reactivation in a cohort of 120-150 patients after allo-HSCT. Moreover, the results will be compared to (i) analysis of leukocyte subpopulations and (ii) multimer techniques detecting CMV-specific CD8 positive T lymphocytes (CTL) (optional).

Demonstrating the suitability of the improved T-Track® CMV assay to identify patients at reduced risk for recurrent CMV-reactivation, CMV disease or GvHD would highly improve and optimize follow-up care after allo-HSCT regarding therapy success as well as reduced public health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving an allogeneic hematopoietic stem cell transplantation being either CMV seropositive or receiving a graft from a CMV seropositive donor or both, donor and recipient are CMV seropositive (D+/R-, D-/R+, D+/R+)
* Patients receiving a first allogeneic hematopoietic stem cell graft
* Patient at least 18 years of age
* Written informed consent

Exclusion Criteria:

* Seronegativity for CMV both for patient and donor (D-/R-)
* Patients receiving standard anti-CMV prophylaxis
* Patients receiving a haploidentical allogeneic hematopoietic stem cell graft
* Patients receiving an umbilical cord blood graft
* Patients treated with Alemtuzumab (e.g. Campath)
* Patient has any form of substance abuse, psychiatric disorder or condition that, in the opinion of the investigator may invalidate communication with the investigator
* Lack or withdrawal of informed consent
* Patient is unable to comply with the visit schedule in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving an allogeneic hematopoietic stem cell transplantation for the first time, being either CMV seropositive or receiving a graft from a CMV seropositive donor or both, donor and recipient are CMV seropositive
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Determination of changes in pp65 and/or IE-1 specific CMI applying T-Track® CMV | days 45, 60 and 80 post Tx as well as at any time between day 45 - 225 in case of CMV-complications

SECONDARY OUTCOMES:
Changes in CMV viral load measured by CMV-PCR | As defined in the respective guidelines of the participating institutes, at least in parallel with T-Track® CMV, any time between day 0 - 225
Determination of frequencies of leukocyte subpopulations | In parallel with T-Track® CMV, thus days 45, 60 and 80 post Tx as well as at any time between day 45 - 225 in case of CMV-complications
  Numbers of naïve (CD45RA) and memory (CD45RO) CD4 and CD8 positive T cells (CD3) as well as NK cells (CD56) and monocytes (CD14) determined by flow cytometry

OTHER OUTCOMES:
Determination of numbers of CMV-specific CTL applying a multimer staining for CMV epitopes | In parallel withT-Track® CMV, thus days 45, 60 and 80 post Tx as well as at any time between day 45 - 225 in case of CMV-complications, optional
Determination of occurrence and severity of GvHD | Any time during study period (day 0 - 225)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Wolff, Prof. Dr. med., Principal Investigator — Klinik für Innere Medizin III, Hämatologie und Onkologie Regensburg
Locations (1):
- Universitätsklinikum Regensburg, Regensburg, Germany

REFERENCES:
- [Derived] Wagner-Drouet E, Teschner D, Wolschke C, Janson D, Schafer-Eckart K, Gartner J, Mielke S, Schreder M, Kobbe G, Kondakci M, Hilgendorf I, von Lilienfeld-Toal M, Klein S, Heidenreich D, Kreil S, Verbeek M, Grass S, Ditschkowski M, Gromke T, Koch M, Lindemann M, Hunig T, Schmidt T, Rascle A, Guldan H, Barabas S, Deml L, Wagner R, Wolff D. Standardized monitoring of cytomegalovirus-specific immunity can improve risk stratification of recurrent cytomegalovirus reactivation after hematopoietic stem cell transplantation. Haematologica. 2021 Feb 1;106(2):363-374. doi: 10.3324/haematol.2019.229252. PMID 31879324
- See also: Lophius Biosciences GmbH — http://lophius.com